CLINICAL TRIAL: NCT07047872
Title: Patient Reported Outcomes Post-Mastectomy and In-house 3D-printed Individualized External Breast Prostheses
Brief Title: A 3D-Printed External Breast Prosthesis for the Improvement of Patient-reported Outcomes Among Breast Cancer Patients That Underwent a Mastectomy Without Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-004692; NCI-2024-10468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-004692 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-06-16; First posted 2025-07-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (3D-printed external breast prosthesis) (Experimental): Patients undergo CT, development of a patient-specific external breast prosthesis model using CAD, and measurements for 3D-printed external breast prosthesis during screening. Patients then undergo fitting for and receive the 3D-printed external breast prosthesis on study.
  Interventions: Procedure: Computer-Aided Diagnosis; Procedure: Prosthetics Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computer-Aided Diagnosis — Undergo CAD development for patient-specific external breast prosthesis model
  Other Names: CAD
Procedure: Prosthetics Intervention — Undergo measurements for external breast prosthesis
Procedure: Prosthetics Intervention — Undergo fitting for 3D-printed external breast prosthesis
Procedure: Prosthetics Intervention — Receive 3D-printed external breast prosthesis
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether a three-dimensional (3D)-printed external breast prosthesis improves patient-reported outcomes (PRO) among breast cancer patients that underwent surgical removal of the breast (mastectomy) without surgical reconstruction. Breast cancer remains a significant health concern and often requires a mastectomy. While breast reconstruction is a common option following a mastectomy, some patients decide not to undergo it or are not candidates. An external breast prosthesis is worn on the outside of the body to replace the breast that was removed during the mastectomy. Traditional external breast prostheses may lack comfort and fit. A 3D-printed external breast prosthesis is customized to the patient using 3D imaging along with computer-aided design (CAD) to interpret the 3D imaging to develop and print a patient-specific external breast prosthesis. This may create a better fitting prosthesis which may improve PRO.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals aged 18 years or older
* History of unilateral or bilateral mastectomy for any indication
* No implant or autologous reconstruction

  * Allowed: Goldilocks closure, flat closure, simple skin closure
* Willingness to participate in the study by completing PRO assessments or receiving personalized 3D-printed breast prostheses
* Ability to provide informed consent
* Ability to complete study procedures, including surface scanning (with temporary fiducial skin markers), standardized photography, and surveys at 1, 3, 6, and 12 months

Exclusion Criteria:

* Individuals with contraindications for participation, such as severe medical conditions that may interfere with study procedures
* Lack of willingness or capacity to provide informed consent for study participation
* Inability to communicate effectively in the study language (e.g., English)
* Patients with open wounds, active infection, or dermatologic conditions at the chest/breast site that would interfere with scanning, fiducial marker placement, or prosthesis use
* Patients unwilling or unable to undergo surface scanning, standardized photography, or complete survey follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
Patient-reported satisfaction with appearance | At baseline, 1 month, 3 months, 6 months, and 1 year
  Will be assessed by patient self-reported satisfaction with appearance and evaluated descriptively.
Patient-reported emotional well-being | At baseline, 1 month, 3 months, 6 months, and 1 year
  Will be assessed by a an Emotional Response survey, which consists of 12 questions answered on a five-point Likert scale ranging from strongly disagree to strongly agree.

SECONDARY OUTCOMES:
Patient-reported comfort of personalized three-dimensional (3D)-printed breast prosthesis | At baseline, 1 month, 3 months, 6 months, and 1 year
  Will be assessed by patient response on a 5-point Likert scale ranging from very dissatisfied to very satisfied.
Patient-reported fit of personalized 3D-printed breast prosthesis | At baseline, 1 month, 3 months, 6 months, and 1 year
  Will be assessed by patient response on a 5-point Likert scale ranging from very dissatisfied to very satisfied.
Patient-reported satisfaction with personalized 3D-printed breast prosthesis | At baseline, 1 month, 3 months, 6 months, and 1 year
  Will be assessed by a Prostheses Evaluation survey, which consists of 11 questions answered on a five-point Likert scale ranging from very dissatisfied to very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Vijayasekaran, MBBS, Principal Investigator — Mayo Clinic; Sandhya Pruthi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials